CLINICAL TRIAL: NCT00002371
Title: A Randomized Double-Blind Study of Safety, Virologic and Immunological Effects of Stavudine Plus Lamivudine (3TC) Versus Zidovudine Plus Lamivudine in HIV-Infected Subjects Following At Least Six Months of Zidovudine Therapy
Brief Title: The Safety and Effectiveness of Lamivudine Plus Stavudine or Zidovudine in HIV-Infected Patients Who Have Taken Zidovudine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 244B; AI455-048
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2011-04

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; Stavudine; Lamivudine; RNA, Viral; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Lamivudine; Stavudine; Zidovudine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Lamivudine
Drug: Stavudine
Drug: Zidovudine

SUMMARY:
To compare the magnitude and durability of the reduction in plasma HIV RNA in the two treatment groups over the first 12 weeks of treatment. To determine the safety of each of the two treatment groups.

DETAILED DESCRIPTION:
Patients will be randomized to either Stavudine (d4T) + Lamivudine (3TC) + Zidovudine placebo or Zidovudine (ZDV) + Lamivudine + Stavudine placebo. Patients whose plasma HIV RNA levels remain >= 500 copies/ml after 8 weeks of blinded double combination therapy will have indinavir added to their treatment regimen at the week 12 visit.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* At least six months of prior cumulative ZDV therapy.
* Qualifying plasma HIV RNA count of >= 4 log10 copies/ml obtained within 2 weeks of randomization.

Exclusion Criteria

Co-existing Condition:

Patients with any of the following symptoms or conditions are excluded:

* Presence of newly diagnosed AIDS defining opportunistic infection requiring acute therapy at time of enrollment.
* Intractable diarrhea (>= 6 loose stools/day for >= 7 consecutive days).
* Signs and symptoms of bilateral peripheral neuropathy >= grade 2 at the time of screening.
* Inability to tolerate oral medication.
* Any other clinical conditions that in the opinion of the investigator, would make the patient unsuitable for study or unable to comply with the dosing requirements.

Concurrent Medication:

Excluded:

* Therapy with agents with systemic myelosuppressive, neurotoxic pancreatotoxic, hepatotoxic or cytotoxic potential.
* Therapy with rifampin, rifabutin, terfenadine, astemizole, cisapride, triazolam, midazolam and ketoconazole at any time while on indinavir therapy.

Patients with any of the following prior conditions or symptoms are excluded:

* History of acute or chronic pancreatitis.
* Prior history of bilateral peripheral neuropathy.
* Intractable diarrhea (>= 6 loose stools/day for >= 7 consecutive days) within 30 days prior to study entry.

Prior Medication:

Excluded:

* Any prior antiretroviral therapy except for ddI, ddC, 3TC or ZDV (for ZDV, as specified in inclusion criteria).
* Previous therapy with agents with significant systemic myelosuppressive, neurotoxic pancreatotoxic, hepatotoxic or cytotoxic potential within 3 months of study start.
* Therapy with rifampin, rifabutin, terfenadine, astemizole, cisapride, triazolam, midazolam and ketoconazole within 2 weeks prior to starting indinavir.
* Any other prior therapy that, in the opinion of the investigator, would make the patient unsuitable for study or unable to comply with the dosing regimen.

Risk Behavior:

Excluded:

* Active alcohol abuse, sufficient in the investigator's opinion, to prevent compliance with study therapy or to increase the risk of developing pancreatitis.

Required:

At least 6 months of prior cumulative ZDV therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 1996-06; Primary Completion 1997-12 (Actual); Study Completion 1997-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (5):
  - Harbor UCLA Med Ctr, Torrance, California
  - Univ of South Florida, Tampa, Florida
  - SUNY at Stony Brook / Division of Infectious Diseases, Stony Brook, New York
  - Houston Clinical Research Network / Div of Montrose Clinic, Houston, Texas
  - Univ of Utah / School of Medicine / Div of Infect Dis, Salt Lake City, Utah
- Canada (2):
  - Sunnybrook Health Science Ctr, North York, Ontario
  - Montreal Gen Hosp / Div of Clin Immuno and Allergy, Montreal, Quebec
- Univ of Puerto Rico School of Medicine, San Juan, Puerto Rico